CLINICAL TRIAL: NCT02972775
Title: 15-year Mortality After Hospitalization for Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: MORTCOP
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Pauline van Hirtum, MD, Zuyderland Medisch Centrum
Other Study IDs: 16N164
Record Dates: First submitted 2016-10-24; First posted 2016-11-23 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Exacerbation Copd; Mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no interventions. observational study

SUMMARY:
The investigators examine the 15-year mortality after an admission for an exacerbation of Chronic Obstructive Pulmonary disease (COPD).

DETAILED DESCRIPTION:
Several prognostic factors will be examined. Cause of death will be examined. Data will be recruited from medical records and calling general practitioners to find out if a patient is still alive. Statistical analysis will be done with Kaplan Meier, Cox proportional hazards and Chi square

ELIGIBILITY:
Inclusion Criteria:

* admission with exacerbation of COPD

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with an exacerbation of Chronic obstructive pulmonary disease in the Zuyderland medical Centre from 1996 - 1999
Sampling Method: Non-Probability Sample
Enrollment: 845 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients that died after 15 years | 15 years
  Mortality after 15 years

SECONDARY OUTCOMES:
Prognostic factors for mortality | 15 years
  Age (years), Gender (M / F), Previous hospitalization in the past year (yes/no), Re-admission in the next 5 years (number of readmissions per year), forced expiratory volume in 1 second (in liter), Hypercapnia (carbon dioxide in arterial blood in stable condition above 5.9 kiloPascal (kPa) or not), TLCO (transfusion capacity of the lung for carbon monoxide in percentage of predicted, ml / min / kPa), Comorbidity (Charlson Comorbidity Index) Date and cause of death
Cause of death | 15 years
  Chronic obstructive pulmonary disease, lung carcinoma, cardiovascular, other

CONTACTS AND LOCATIONS:
Overall Officials: Martijn de Kruif, MD, PhD, Principal Investigator — Zuyderland Medical Center
Locations (1):
- Zuyderland Medical Center, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Traver GA, Cline MG, Burrows B. Predictors of mortality in chronic obstructive pulmonary disease. A 15-year follow-up study. Am Rev Respir Dis. 1979 Jun;119(6):895-902. doi: 10.1164/arrd.1979.119.6.895. PMID 453709